CLINICAL TRIAL: NCT02431182
Title: Randomized Control Trial to Evaluate the Effectiveness of Memory Training Workshops in People From 65 to 80 Years
Brief Title: Trial to Evaluate the Effectiveness of Memory Training Workshops in People From 65 to 80 Years
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI11/02060
Record Dates: First submitted 2015-04-22; First posted 2015-04-30 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2014-12

CONDITIONS: Memory Loss; Age-Related Memory Disorders
MeSH Terms: conditions — Memory Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Memory training group (Experimental): Memory training:The intervention consists of twelve 90-minutes group sessions given once a week by a specialized psychologist.
  The groups are formed by around 15 people. Each session has its own objectives, material and activities. The content of the intervention is based on memory training from different perspectives as cognitive and emotional aspects or social and individual skills.
  Interventions: Behavioral: Memory Training Workshop
- Control group (No Intervention): No intervention will be administred until the delayed post-test is finished

INTERVENTIONS:
Behavioral: Memory Training Workshop — 1. Presentation of the workshop: Objectives and Methodology
  2. Explanation of the different types of memory and its implication in normal life
  3. Strategies for gathering and codification of the information
  4. Strategies for selection and storage the information
  5. Strategies for gathering, codification, selection, storage and recuperation of the information. Importance of the context and the meaning of things. Semantic and episodic memory
  6. Strategies for gathering, codification, selection, storage and recuperation of the information. Individual differences
  7. Strategies for recuperation according to the individual profile. Improving self-esteem
  8. Strategies for recuperation Social skills.
  9. Personal and social skills
  10. New contexts and opportunities
  11. Evaluation of the workshop
  Arms: Memory training group

SUMMARY:
Randomized controlled trial to assess the effectiveness of a Memory Training Workshop in cognitive function, in terms of self-perceived memory, everyday memory and executive control abilities. It is expected that the group intervention of memory training that this study proposes significantly improves cognition (memory, attention and executive control abilities) and the quality of life related to health (HRQOL) in the Experimental Group (EG) compared to the Control Group (CG). The group of individuals that take part in the Memory Training Workshops (Experimental Group) will be compared to another group of similar characteristics that do not (Control Group). Data will be collected at baseline, 3 months later and 6 months later.

DETAILED DESCRIPTION:
Study design: Randomized controlled trial, comparing one group of individuals that take part in the Memory Training Workshops (Experimental Group) with another group of similar characteristics that do not (Control Group). Data will be collected at baseline, 3 months later and 6 months later.

Setting: The study will be done in Health Care Centres of Barcelona City (Spain) Randomization unit: Individuals Study Population: Healthy older people belonging to the four Health Care Centres included in the study and that meet the inclusion criteria

Description of the study procedure:

1. Recruitment and screening: Recruitment will be conducted in the four participating Health Care Centres through printed materials.(leaflets and posters) in the Health Care Centres and close community sites (library, pharmacy, market or elderly meeting centre). Interested individuals will have to contact their corresponding Health Care Centre where they will be first screened regarding age (older than 65 and younger than 81) and previous memory training (not having been involved in memory training during the 3 previous years). Those who meet both criteria will be cited for a inclusion interview with a study-trained doctor or nurse at the Health Care Centre.
2. Inclusion and randomisation: Informed consent follows the requirements of the institution's Ethics Comitee. Written consent to participate will be obtained in-person assessment at the beginning of the screening interview. Selection of the participants will be performed through the screening interview, where data will be sought for regarding socio-demographic questions, the Short version of the Geriatric Depression Scale (GDS-5), the Mini Mental State Examination (MMSE) and the medical history with the active clinical diagnoses and active medication. After the screening interview and if the participant is eligible and willing, the individual will be randomly assigned to the EG or to the CG through a closed and opaque envelope with the group information inside. Total time required for screening is around 30 minutes.
3. Baseline and follow-up assessments: Three assessments will be conducted through the study: at baseline after randomisation, post-intervention at time-point between 3 and 4 months post-baseline (immediate post-test), follow-up at time-point 6 months post-baseline (delayed post-test). All three assessments will collect information on variables detailed in Table 1, and will be conducted by a trained psychologist trough in-person interviews in the Health Care Centre. Time requirements will be around 75 minutes for the baseline assessment, and around 90 minutes for the follow-up assessments
4. Implementation of the intervention by the experimental group: Once the baseline assessment is conducted, the individuals of the EG will start the multifactorial intervention. The memory training workshop is designed to stop or delay memory losses age-related and to promote personal autonomy enhancing mental and physical wellbeing. Concretely, it pretends to wider the knowledge about memory function, to improve memory process and to increase self-esteem and the quality of life by giving some strategies and some relational space. The intervention consists of twelve 90-minutes group sessions given once a week by a specialized psychologist. The groups are formed by around 15 people. Each session has its own objectives, material and activities. The content of the intervention is based on memory training from different perspectives as cognitive and emotional aspects or social and individual skills.
5. Standardization of Assessment: Standardization of data collection procedures will be ensured through a variety of training and quality-control procedures. Data collectors will be masked with regard to treatment group assignment. All data collectors will participate in an intensive 2-day training workshop which includes information about the study design, recruitment issues, and general research interviewing principles; detailed instruction in the administration of each test or measurement procedure; demonstrations of each test/measurement; and practice sessions with other data collectors. Furthermore, they will use an easy and friendly answer sheet specially designed for the study. Fulfilled sheets will be always reviewed by the fieldwork coordinator, who in case of missing data or possible mistakes will contact with data collectors to solve any doubt.

ELIGIBILITY:
Inclusion Criteria:

* People of both sexes between 65 and 80 years old (including these ages) who consent to participate in the study.
* Not presenting diagnoses of dementia or cognitive impairment measured through the Mini-Mental State Examination (MMSE >24)
* Absence of depression measured by the Geriatric Depression Scale (GDS 5 ≤ 2)

Exclusion Criteria:

* Having participated in a memory training within the last 3 years
* Having a severe sensorial disability
* Being illiterate/can not read or write

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 300 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Everyday Memory at 3 and 6 months measured by the Rivermead Behavioural Memory test | baseline, at 3 months from baseline and at 6 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Anna Pérez, MPH, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Agència de Salut Pública de Barcelona, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Perez A, Roque M, Domenech S, Monteserin R, Soriano N, Blancafort X, Bosom M, Vidal C, Petit M, Hortal N, Gil C, Espelt A, Lopez MJ. Efficacy of memory training in healthy community-dwelling older people: study protocol for a randomized controlled trial. BMC Geriatr. 2015 Oct 1;15:113. doi: 10.1186/s12877-015-0110-4. PMID 26429559